CLINICAL TRIAL: NCT02149862
Title: FIRBladd - Use of Infrared Spectroscopy in the Diagnosis of Bladder Tumors
Acronym: FIRBladd
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-A00038-37
Record Dates: First submitted 2014-05-13; First posted 2014-05-29 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2014-05

CONDITIONS: Bladder Cancer
Keywords: Bladder cancer; Diagnostic; Infrared; Spectrum; Urina; Patients with an indication of partial or total bladder resection; or; Lithiasic patients should be operated a urinary calculation, without catheter "double J"
MeSH Terms: conditions — Urinary Bladder Neoplasms; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cancer (Experimental): patients with an indication of partial or total bladder resection will have urine infrared analysis
  Interventions: Other: Urine infrared analysis
- control group (Placebo Comparator): Lithiasic patients should be operated a urinary calculation, without catheter "double J", will have urine infrared analysis
  Interventions: Other: Urine infrared analysis

INTERVENTIONS:
Other: Urine infrared analysis — Collected urine sample will be stored at -80°C for further infrared analysis. Spectra will be analyzed by visual inspection, and statistical method such as Principal Components Analysis and logistic regressions methods.

SUMMARY:
The purpose of this study is too assess infrared spectroscopy ability to discriminate urine of a patient affected by bladder cancer from urine of reference patient.

DETAILED DESCRIPTION:
Bladder Cancer is the ninth cause of cancer worldwide, and it is still developing, due to growing risk factors such as Tobacco consumption. It has a high level of recurrence, which imposes regular screening and permanent treatment to the patient that has developed a bladder tumor.

Bladder cancer main symptom is blood in the urine, which has low specificity and sensibility. Other screening methods include cytology and image through cystoscopy. Conclusive diagnostic is performed by biopsy of the suspicious lesions. The latter methods are highly invasive.

Hence, it is necessary to develop non invasive technique for bladder cancer screening and follow up, as there is no reliable prognostic factor available. The investigators expect to improve the detection level in the urine by measuring and analyzing its absorption spectrum in the mid infrared, spectrum which provides a comprehensive image of metabolic situation.

Hence, the main objective of the study is to assess infrared spectroscopy ability to discriminate urine of a patient affected by bladder cancer from urine of reference patient. Success will be evaluated upon the discrimination level of cancer affected patient urine infrared spectrum vs. standard patient ones.

Secondary objective will be to assess the capability to detect different affection levels and tumors grade through the infrared spectrum analysis, as well as the predictive potential of the technique. The investigators may also assess the test intrinsic sensibility and specificity.

The study is planned over an 18 month period of time, to collect urine from 100 patients followed up at Rennes Hospital center for bladder cancer treatment and from a reference pool of 100 patients cured for kidney stones. All donors will be cognizant volunteers, adult from both genders. Minors, pregnant or breast feeding women, protected adults, patients also treated for other cancers, or the ones treat with a "double J" probe will not be included into the study.

Clinical data will be extracted out of patient file (sex, age, weight, size and resected tumor characteristics).

Collected urines will be submitted to the standard cytologic analysis. Resected tumors will be analyzed by Rennes hospital anatomic pathology laboratory according to standard procedure.

Collected urine sample will be stored at -80°C for further infrared analysis.

As this is a preliminary study, there is no existing data to calculate the size of a statistically relevant sample.

Hence, the investigators chose to include 100 patients of each category to fit with Rennes hospital capacities during the time of the study.

Spectra will be analyzed by visual inspection, and statistical method such as Principal Components Analysis and logistic regressions methods.

This model will allow to determine spectral area with discriminating values between both populations. The wavelength of these spectral areas will be eventually correlated to biological elements absorption to confirm their relevance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an indication of partial or total bladder resection
* Lithiasic patients should be operated to a urinary calculation, without catheter "double J"
* Free inform and written consent

Exclusion Criteria:

* Patients also treated for other cancers
* Lithiasic patients with catether "double J"
* Pregnant or breast feeding women
* Protected adults,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
infrared spectroscopy | the measure will be realized at the end of the studie, an expected average 18 month after the first inclusion
  14 bands with a major local optimum value is retained on the spectrum. For each band, the positions and intensities of local optima are the set of explanatory variables. Discriminating threshold is estimated by validation Cross and chosen to have the best compromise between sensitivity and specificity.

SECONDARY OUTCOMES:
TNM system (tumor-nodes-metastasis) | the classification of the operating room will be carried out the day of the intervention or approximately 8 weeks after the inclusion
  Resected tumors will be analyzed by Rennes hospital anatomic pathology laboratory according to standard procedure

CONTACTS AND LOCATIONS:
Overall Officials: Karim KB Bensalah, PU-PH, Principal Investigator — CHU Rennes
Locations (1):
- CHU rennes, Rennes, France